CLINICAL TRIAL: NCT06323850
Title: Improving Access to Community-Based Occupations Via a Rideshare Training Progra
Brief Title: Improving Access to Community-Based Occupations Via a Rideshare Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Organization for Autism Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20028878
Record Dates: First submitted 2024-02-06; First posted 2024-03-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Autism
Keywords: Community Mobility; Rideshare
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Single group, pre- and post-test. Subjects were measured 8 times during intervention stage and 8 times during the follow-up stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): The experimental group will receive the intervention then a 2-month follow-up
  Interventions: Behavioral: Intervention Phase; Behavioral: Virtual Training Sessions; Behavioral: Ride-Along Training Sessions

INTERVENTIONS:
Behavioral: Intervention Phase — After participants have been enrolled, they will be assigned to one of the trainer-pairs and will work with them to schedule the first two sessions. Most clients will be able to schedule one virtual session per week and one ride along session per week for the first five weeks, with the remaining three weeks allotted to practice ride-along sessions and module repetition (as needed). The additional time also provides a buffer if subjects are unavailable for a week during the intervention phase.
Behavioral: Virtual Training Sessions — Virtual sessions will take place over Zoom each session lasting 20-30 minutes. Each of the five virtual sessions will be aligned with the five online modules. For each module, exercises are built in to test comprehension. If the participant does not complete an exercise accurately, the lead trainer will explain why the response was incorrect and prompt them to repeat the video modeling exercise. The support training partner will take notes to support the formative assessment process and complete fidelity checks.
Behavioral: Ride-Along Training Sessions — The first ride-along session will be the baseline session for assessing level of independence (number of cues needed) and safety. The participant will have up to 8 ride-along sessions to reach full independence (no cues needed) and full marks on the safety assessment. The lead trainer will provide the cues as needed to complete each step of the Rideshare process.

SUMMARY:
Community mobility is critical for living independently and engaging in one's community. It is especially important for people in their early adult years, as this is often a time of transition to employment and living independently. Community mobility can be particularly challenging for adults with Autism Spectrum Disorders (ASD) (henceforth referred to as autistic adults based on the preferred identity-first language of our autistic partners). Some autistic adults are unable to meet the demands of driving. Public transportation is an option for autistic adults; and autistic adults are more likely to use public transportation than their non-autistic counterparts. However, using public transportation may be just as challenging as driving for the autistic population. Rideshare (also called ride-hailing) is a relatively new form of transportation in which passengers get from point A to point B in private vehicles driven by their owners. A digital app, usually accessed on a smartphone, matches passengers and drivers, coordinates routes using a GPS system, and facilitates payment through a linked financial account. Rideshare has the potential to address many of the issues autistic adults have accessing the community. It is faster and more direct than the public train or bus, there is limited social interaction required, and rides can be scheduled at any time. Despite it's potential to increase transportation in autistic adults, there are no evidence-based training programs to support Rideshare use in this population.

DETAILED DESCRIPTION:
Rideshare services are widely adopted across the globe and provide a safer, more flexible, and less taxing transportation option for many individuals. Rideshare can help people to get to more places they want to go and allows for spontaneity since a ride can be arranged in the moment, at any time of day. Rideshare picks passengers up and drops them off at their specific destination, eliminating the need to walk to bus stops, wait at stations, or transfer to more than one bus or train. Not only does this save time, it may increase safety especially at night or during inclement weather. Rideshare may also be more reliable for getting to work on time. Finally, while communicating with the driver may be a challenge, there is only one person with which to interact versus potentially many people waiting at stations or on the bus or train.

While the use of Rideshare has the potential to improve community access and expand occupational engagement for autistic adults, few training resources exist to introduce clients to this mode of transportation, assess readiness, or build confidence. Our Rideshare training program has proven feasible to conduct with autistic adults living in an urban-based semi-structured independent housing residence. This study will test the effectiveness and implementation of the SRP program in a wider range of autistic adults living in the central Virginia region

ELIGIBILITY:
Inclusion Criteria:

* study participants have to be 18+ years of age
* living within 100 miles of Richmond, Virginia
* Participants have to have diagnosis of ASD given by a licensed medical professional.
* Participants need to have a stable internet connection
* ability to communicate independently (verbally or via alternative communication device) in English
* have the motoric skills needed to independently use a smartphone (fine motor) and get in and out of a car (gross motor).
* Participants must own a smartphone and be familiar with texting and/or email.

Exclusion Criteria:

* participants who have a severe or profound intellectual disability (IQ below 35) given that the training was designed for those with moderate IQ and above with the potential to travel alone to familiar places
* exclude any individual who already uses Rideshare independently.
* exclude pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Evaluate autistic adults participating in the SRP intervention find the intervention acceptable? | Baseline and after phase 1 (5 weeks)
  Autistic adults participating in the SRP will rate 75% of the items on the Acceptability Intervention Measure (AIM) as Agree or Completely Agree. The AIM is a 5-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Acceptability refers to determining how well an intervention will be received by the target population and the extent to which the new intervention or its components might meet the needs of the target population and organizational setting.
Evaluate if the trainers conducting the SRP intervention find the intervention to be appropriate | Baseline and after phase 1 (5 weeks)
  Trainers conducting the SRP intervention will rate 75% of the items on the Intervention Appropriateness Measure (IAM) as Agree or Completely Agree. The AIM is a 5-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Acceptability refers to determining how well an intervention will be received by the target population and the extent to which the new intervention or its components might meet the needs of the target population and organizational setting.
Autistic adults who have participated in the SRP program display greater independence in using Rideshare | Baseline and after phase 1 (5 weeks)
  Autistic adult who have participated in the SRP program will display greater independence in using Rideshare
Autistic adults who have participated in the SRP program display greater safety in using Rideshare | Baseline and after phase 1 (5 weeks)
  Autistic adult who have participated in the SRP program will display greater safety when using Rideshare

SECONDARY OUTCOMES:
How do SRP participants use of Rideshare for community, social, and/or employment activities after the intervention | Baseline and after phase 1 (5 weeks) and 3 months post intervention
  This is an exploratory research question and the investigators will use descriptive statistics and visual analyses to look at trends in how Rideshare is used after participation in the SRP program. The investigators will also gather qualitative data through post-intervention interviews with participants to help determine the impact of the program and what improvements are needed.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Reynolds, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States